CLINICAL TRIAL: NCT07135323
Title: AvertD Post-Approval Study
Status: Recruiting | Type: Observational
Sponsor: Prescient Medicine Holdings, Inc. (Industry)
Collaborators: Caron Treatment Centers (Other); Concentrics Research (Other)
Responsible Party: Sponsor
Other Study IDs: TP-60418
Record Dates: First submitted 2025-07-17; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Genetic: Opioid Used Disorder Risk Assessment — Determine the likelihood of Opioid Used Disorder prior to prescribing opioids

SUMMARY:
A Prospective Post-Approval Study of AvertD to Evaluate Device Performance, Prescribing Impact, and Labeling Comprehension in the Intended Use Population

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Prior to first opioid prescription
* Being considered for first oral opioid prescription (4-30 days)
* Prescribed AvertD as part of care
* Willing and able to complete yearly assessments for 5 years
* Signed informed consent

Exclusion Criteria:

* Planned opioid prescription <4 or >30 days
* Any condition making participation unsafe or infeasible per investigator judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects being considered for first oral opioid prescription (4-30 days)
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of AvertD | Measured over 5 years
  Comparison of Averted results to diagnosis of Opioid Used Disorder from M.I.N.I. tool

CONTACTS AND LOCATIONS:
Locations (1):
- Concentrics Research, Indianapolis, Indiana, United States